CLINICAL TRIAL: NCT06770829
Title: The Effect of a Preventive Diabetic Foot Care Program on Knowledge, Behavior, Self-Management, and Glycemic Control Levels in Patients at Risk of Diabetic Foot
Brief Title: Implementation of a Preventive Diabetic Foot Care Program for Patients at Risk of Diabetic Foot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sultan Patat, MSc, Lecturer, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Akdeniz U3820
Record Dates: First submitted 2024-12-04; First posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Foot Ulcer; Type 2 Diabetes Mellitus With Complication
Keywords: Nursing; Type 2 Diabetes Mellitus; Diabetic Foot; Preventive Diabetic Foot Care; Randomized Controlled Trial
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2 | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The DiaFOOTCare Program evaluates its impact on knowledge, behavior, self-management, and glycemic control by randomizing 78 type 2 diabetes patients with diabetic foot risk into intervention (n = 39) and control (n = 39) groups using block randomization (1:1 ratio). The intervention group receives educational tools, including an e-booklet with voice-over modules, a foot care checklist, a training video, a 20-25-minute face-to-face session, and personalized goal-tracking cards to monitor progress over three months. SMS reminders are sent three times weekly, and materials are shared via WhatsApp or email for accessibility. The control group receives a Ministry of Health brochure on diabetic foot care, explained using a tablet, and the same goal-tracking card as the intervention group. Post-intervention assessments, including diabetic foot knowledge, behavior, self-management scales, glycemic control, and goal card reviews, will determine program effectiveness after three months.
Who Masked: Participant
Masking Description: Participants will be assigned to groups based on a randomization list created to ensure balanced allocation. The assignment of participants to the intervention and control groups, as well as the evaluation of outcome measurement data, will be conducted by two independent investigators.
  Although the researchers delivering the interventions will not be blinded to group assignments, participant blinding will be maintained. Participants will remain unaware of the study hypotheses and the group to which they have been assigned, ensuring that their responses and engagement are not influenced by this knowledge.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DiaFOOTCare Group (Experimental): The DiaFOOTCare Group will receive interventions to support diabetic foot self-management. An e-booklet on type 2 diabetes management and preventive diabetic foot care will be shared via WhatsApp or email, along with audio modules for easy access. An educational video featuring a simulated patient will demonstrate preventive foot care practices and be shared digitally. A 25-30-minute face-to-face training session will provide personalized guidance using a tablet. Goal-tracking cards will establish three-month behavioral goals, with patients documenting progress. SMS reminders will be sent three times weekly to reinforce adherence. Patients will have access to DiaFOOTCare resources for 12 weeks. At the three-month follow-up, outcomes will be assessed using the Glycemic Control Form, Goal-Tracking Card, Diabetic Foot Knowledge Scale, Foot Care Behavior Scale, Nottingham Functional Foot Care Diagnostic Form, and Diabetic Foot Self-Management Scale.
  Interventions: Behavioral: DiaFOOTCare Program
- Active Control Group (Active Comparator): The active control group will receive routine outpatient follow-ups and a diabetic foot care brochure from the Ministry of Health, explained by the researcher and shared via WhatsApp or email. Goal-tracking cards from the DiaFOOTCare program will be used to set individual diabetic foot self-management behavioral goals collaboratively during the initial interview. Patients will be instructed on how to complete the cards and maintain them over a three-month period. Post-tests will be conducted at the three-month follow-up to evaluate outcomes using the Glycemic Control Form, Goal-Tracking Card, Diabetic Foot Knowledge Scale, Foot Care Behavior Scale, Nottingham Functional Foot Care Diagnostic Form, Diabetic Foot Development Follow-up Form, and Diabetic Foot Self-Management Scale. After the follow-up, the e-booklet, audio modules, and preventive foot care video from DiaFOOTCare will be shared via WhatsApp or email to provide additional education and support.
  Interventions: Behavioral: Ministry of Health and Education

INTERVENTIONS:
Behavioral: DiaFOOTCare Program — The DiaFOOTCare Program includes initiatives to support diabetic foot self-management. An e-booklet on type 2 diabetes management and preventive foot care will be shared via WhatsApp or email, along with audio modules for convenient access. An interactive video featuring a simulated patient will visually demonstrate preventive foot care practices and will also be shared digitally. A 25-30-minute face-to-face training session will provide personalized education using a tablet. Goal-tracking cards will be introduced to collaboratively set three-month behavioral goals, with patients documenting their progress during the follow-up. SMS reminders will be sent three times weekly to reinforce adherence. Patients will have digital access to all DiaFOOTCare resources, including the e-booklet, audio modules, and video, for 12 weeks, ensuring accessibility via WhatsApp or email. These measures aim to enhance knowledge, behavior, and self-management practices in preventive diabetic foot care.
  Other Names: Ministry of Health and Education
  Arms: DiaFOOTCare Group
Behavioral: Ministry of Health and Education — The active control group will receive routine outpatient follow-ups and a diabetic foot care brochure from the Ministry of Health, explained by the researcher and shared via WhatsApp or email for reference. Goal-tracking cards from the DiaFOOTCare program will be used to set individual diabetic foot self-management behavioral goals collaboratively during the initial interview. Patients will be instructed on how to complete the cards and maintain them over a three-month period. At the end of the follow-up, post-tests will assess outcomes using the Glycemic Control Form, Goal-Tracking Card, Diabetic Foot Knowledge Scale, Foot Care Behavior Scale, Nottingham Functional Foot Care Diagnostic Form, Diabetic Foot Development Follow-up Form, and Diabetic Foot Self-Management Scale. Educational resources, including the e-booklet, audio modules, and video developed in DiaFOOTCare, will also be shared via WhatsApp or email to provide additional support and enhance diabetic foot self-management.
  Arms: Active Control Group

SUMMARY:
This study aims to evaluate the effect of a preventive diabetic foot care program on the knowledge, behavior, self-management, and glycemic control levels of type 2 diabetic patients at risk of diabetic foot. The development of a Preventive Diabetic Foot Care Program (DiaFOOTCare) for patients with type 2 diabetes at risk of diabetic foot is expected to make a significant contribution to preventing diabetic foot formation. The DiaFOOTCare program consists of two stages. In the first phase, a comprehensive, multi-component, and evidence-based preventive diabetic foot care program will be designed specifically for type 2 diabetic patients at risk of diabetic foot. The internal validity of the program will be tested through expert evaluations by specialists in diabetic foot care, assessments using readability formulas, and pre-application testing with patients identified as being at risk of diabetic foot. As part of the final implementation of the first phase, all interventions included in the DiaFOOTCare protocol will be administered to four patients with diabetic foot risk over a three-week period. Following this, the DiaFOOTCare protocol will be evaluated based on the feedback provided by these four pre-application participants. In the second phase, a randomized controlled trial (RCT) with a single-blinded and active control group design will be conducted at the Akdeniz University Hospital Endocrinology and Metabolic Diseases Outpatient Clinic. A group of patients with type 2 diabetes and diabetic foot risk will be identified, and pre-tests will be administered. The patients will then be randomly assigned to the intervention group (n=39) and the control group (n=39). The effectiveness of the DiaFOOTCare program will be assessed through post-tests.

DETAILED DESCRIPTION:
Diabetic foot, a complication of diabetes, is a significant cause of morbidity and mortality, as well as associated challenges such as high healthcare costs and reduced quality of life. Studies have shown that adherence to treatment among individuals at risk for diabetic foot is consistently low. However, patient education and proper guidance on care can significantly reduce the incidence of foot ulcers. This study aims to evaluate the effect of a preventive diabetic foot care program on the knowledge, behavior, self-management, and glycemic control levels of type 2 diabetic patients with diabetic foot risk. The development of the Preventive Diabetic Foot Care Program (DiaFOOTCare) for patients with type 2 diabetes at risk of diabetic foot is expected to play a pivotal role in preventing diabetic foot formation.

Study Design and Methods This study is structured in two phases. In the first phase, the DiaFOOTCare program will be developed, and in the second phase, its effectiveness will be tested through a randomized active-controlled trial.

First Phase: Development of the DiaFOOTCare Program

The DiaFOOTCare program includes various educational and behavioral interventions:

An e-booklet on type 2 diabetes management and preventive diabetic foot care will be prepared. The e-booklet's content will be recorded as voice-over modules, allowing patients to listen to the training at any time during the follow-up period.

A preventive diabetic foot care checklist will be developed to improve patients' knowledge and behaviors related to foot care, accompanied by a training video featuring a simulated patient.

A 20-25 minute face-to-face training session on preventive diabetic foot care will be provided.

A goal-tracking card will be created to enhance diabetes self-management. During the initial interview, three-month individual diabetes management goals will be collaboratively set with the patients and recorded on their tracking cards. Patients will be instructed on how to complete these cards and will be asked to maintain them throughout the three-month period.

To support patients in achieving their diabetes management goals, Short Message Service (SMS) reminder messages will be sent three times a week. The e-booklet, voice-over modules, and video will be shared via WhatsApp or email, ensuring patients can access these materials on their phones or computers.

Second Phase: Testing the DiaFOOTCare Program The second phase will use a randomized controlled trial (RCT) design with single-blinding and an active control group. This phase will be conducted with type 2 diabetic patients at risk for diabetic foot who are treated at the Akdeniz University Hospital Endocrinology and Metabolism Polyclinic and meet the inclusion criteria.

Participants will be stratified based on their diabetic foot risk (categories 2 and 3 of the International Working Group on the Diabetic Foot [IWGDF] Risk Classification System) and randomized into two groups using stratified block randomization.

The intervention group (n=39) will receive routine outpatient follow-up along with all components of the DiaFOOTCare program over a three-month period.

The active control group (n=39) will be provided with a brochure on preventive diabetic foot care (available from the Ministry of Health website), explained by the researcher, and shared via WhatsApp or email. The control group will also use the goal-tracking card developed within the DiaFOOTCare program.

Outcome Measures At the end of the three-month period, diabetic foot knowledge, behavior, and self-management scales will be administered to all participants as part of the post-test. Glycemic control will be assessed, and the goal-tracking cards completed by the patients will be evaluated.

Sample Size and Randomization The sample size was calculated using the G*POWER software based on an 80% power and a 5% significance level. A total of 78 participants will be included in the study, with 39 patients in each group.

To minimize assignment bias, stratified block randomization will be conducted using an independent researcher not involved in the study. This researcher will use a computer-based randomization method to assign participants to groups and will place the group assignments in opaque envelopes for use during the study. By implementing this method, potential bias during the randomization process is effectively controlled.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria to be included in the study:

* Patients with type 2 diabetes receiving follow-up and treatment at the Akdeniz University Hospital Endocrinology and Metabolic Diseases Outpatient Clinic.
* Presence of one or more diabetic foot risk factors, categorized as category 2 or 3 according to the IWGDF (International Working Group on the Diabetic Foot) Risk Classification System.
* Diagnosed with type 2 diabetes for at least six months.
* Aged between 30 and 65 years.
* Literate.
* No physical or mental disabilities that would prevent answering the study questions.
* No communication barriers.
* Able to understand and verbalize their diagnosis.
* HbA1c ≥7.5%.
* Internet access at home and possession of a device such as a computer, tablet, or smartphone, with the ability to use these tools.
* Willing to provide informed consent to participate in the study.

Exclusion Criteria

Participants will be excluded if they meet any of the following conditions:

* Myocardial infarction, stroke, heart failure, or angina pectoris within the last year.
* Diagnosed with type 1 diabetes or gestational diabetes.
* Presence of an active diabetic foot ulcer.
* Diagnosed with dementia or cognitive deficits.
* Diagnosed with glaucoma, cataracts, or retinopathy.
* Diagnosed with a terminal illness.
* Inability to provide accurate information or participate in the study.

Criteria for Exclusion During Follow-Up

Participants will be excluded from the study during the follow-up period if they meet any of the following conditions:

* Voluntarily choose to withdraw from the study.
* Fail to complete at least two-thirds of the follow-up period for any reason.
* Undergo bariatric surgery during the study.
* Exhibit non-adherence to prescribed medications.
* Have a general health condition that, according to their own statement, is unsuitable for continuing the study.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Diabetes Foot Knowledge Scale | 12 weeks
  The Diabetic Foot Knowledge Scale is a validated tool designed to assess individuals' knowledge of diabetic foot care and complications. It evaluates key areas such as risk factors, preventive strategies, warning signs, and footwear selection. The scale typically includes 20 items, with each correct response earning 1 point, resulting in a score range of 0 to 20. Higher scores indicate strong awareness and reduced risk of complications, while lower scores highlight knowledge gaps requiring targeted education. Psychometric properties include a Cronbach's alpha of 0.63, indicating acceptable internal consistency, and an intra-item correlation coefficient of 0.25. The scale is widely used in clinical and research settings to identify at-risk patients, evaluate educational interventions, and guide strategies to improve diabetic foot self-management. Its practical design makes it a valuable resource for promoting preventive care and reducing diabetic foot complications.
Diabetic Foot Behaviour Scale | 12 weeks
  The Diabetic Foot Behavior Scale is a tool designed to evaluate foot self-care behaviors in individuals with diabetes. The scale consists of 15 items within a single dimension, utilizing a 5-point Likert-type format with responses scored as "Never," "Occasionally," "Sometimes," "Often," and "Always." Total scores range from a minimum of 15 to a maximum of 75, with higher scores indicating better self-care behaviors. The scale has demonstrated good internal consistency, with a reported Cronbach's alpha of 0.83.
Nottingham Functional Foot Care Diagnosis Form | 12 weeks
  The Nottingham Functional Foot Care Diagnosis Form is a comprehensive tool designed to assess foot care practices and identify areas for improvement in individuals with diabetes or other conditions affecting foot health. The form evaluates multiple aspects of foot care through subscales, including hygiene and skin care, nail care, footwear, inspection and monitoring, and symptom management. Responses are scored using a numerical system, often based on frequency or quality of behaviors, with higher scores indicating better foot care practices and lower scores highlighting areas needing improvement or intervention. The form has demonstrated excellent reliability and validity, with Cronbach's alpha values ranging from 0.80 to 0.90, confirming its strong internal consistency.
Diabetic Foot Self-Management Scale | 12 weeks
  The Diabetic Foot Self-Management Scale is a validated tool designed to evaluate self-management behaviors related to diabetic foot care and their impact on glycemic control in patients with diabetes. The scale comprises 16 items that assess various aspects of self-care, including regular foot inspections, appropriate footwear selection, and management of foot-related symptoms. Each item is scored on a Likert-type scale, typically ranging from 1 (never) to 5 (always), resulting in a total score range from 16 to 80. Higher scores indicate better adherence to diabetic foot self-management practices, reflecting a proactive approach to preventing complications such as ulcers or infections. The scale has demonstrated strong reliability, with a reported Cronbach's alpha of 0.85, indicating excellent internal consistency.
Diabetic Foot Development Monitoring Form | 12 weeks
  The Diabetic Foot Evaluation Form is a comprehensive tool used to assess foot health and identify risks for complications in individuals with diabetes. It evaluates key areas such as skin integrity, presence of ulcers or calluses, vascular health, neurological status, and footwear suitability. The form includes both objective clinical assessments and patient-reported inputs, ensuring a thorough evaluation of foot health. The scoring system typically assigns points to various categories, with a higher cumulative score indicating better foot health and lower scores reflecting higher risk levels or areas requiring intervention. For example, scores might range from 0 to 100, where 90-100 represents excellent foot health, 70-89 indicates moderate risk, and below 70 highlights high-risk patients requiring immediate attention. The form has demonstrated strong reliability, with Cronbach's alpha values ranging from 0.80 to 0.90, indicating excellent internal consistency across its components.
Glycaemic Control Form | 12 weeks
  The Glycemic Control Form will be used to evaluate and monitor patients' glycemic control through the analysis of key parameters. These include fasting blood glucose levels (mmol/L), postprandial blood glucose levels (mmol/L), and HbA1c levels (percentage). Fasting and postprandial glucose levels provide immediate insights into daily glucose management, while HbA1c reflects average blood glucose levels over the past 2-3 months, offering a comprehensive picture of long-term glycemic control. These metrics will guide the assessment of patients' diabetes management and inform necessary interventions.
Target Tracking Cards | 12 weeks
  As part of the DiaFOOTCare program, patient goal-tracking cards have been developed to support effective self-management of type 2 diabetes. These cards will facilitate the creation of a three-month individualized goal plan in collaboration with each patient, focusing on adherence to treatment and self-management behaviors. Goals will be set in key areas, including medication adherence, dietary compliance, physical activity, blood glucose regulation, and HbA1c targets. The cards will also document patients' self-reported progress, enabling regular monitoring and adjustment of goals based on their experiences and outcomes. At the end of the three-month period, the information recorded on the goal-tracking cards will be used to evaluate the patient's level of goal achievement and overall progress. This approach ensures a patient-centered, self-report-based method for assessing adherence and facilitating continuous improvement in diabetes management.

CONTACTS AND LOCATIONS:
Overall Officials: Sultan Akcimen Patat, Study Chair — Akdeniz University

IPD SHARING:
Plan to Share IPD: No
This can be shared privately if other researchers wish to obtain it.